CLINICAL TRIAL: NCT03436316
Title: A Phase 1 Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD8154 Following Single and Multiple Ascending Dose Administration in Healthy Subjects.
Brief Title: A Study to Evaluate the Safety, Tolerability and Absorption to the Blood After Administration of Single and Multiple Doses of AZD8154 in Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: D8900C00001
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-07

CONDITIONS: Asthma
Keywords: Phosphoinositide 3-kinase (PI3K) inhibitor; First-in-human (FiH) study
MeSH Terms: conditions — Asthma; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part 1 of this study will be single-blind. Part 2 of this study will be open-label. Part 3 of this study will be single-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- SAD Cohort 1 (Part 1) (Experimental): 6 Participants will receive AZD8154 (single inhaled small particle dose 1) and 2 participants will receive placebo.
  Interventions: Drug: AZD8154
- SAD Cohort 2 (Part 1) (Experimental): 6 Participants will receive AZD8154 (single inhaled small particle dose 2) and 2 participants will receive placebo.
  Interventions: Drug: AZD8154
- SAD Cohort 3 (Part 1) (Experimental): 6 Participants will receive AZD8154 (single inhaled small particle dose 3) and 2 participants will receive placebo.
  Interventions: Drug: AZD8154
- SAD Cohort 4 (Part 1) (Experimental): 6 Participants will receive AZD8154 (single inhaled small particle dose 4) and 2 participants will receive placebo.
  Interventions: Drug: AZD8154
- SAD Cohort 5 (Part 1) (Experimental): 6 Participants will receive AZD8154 (single inhaled small particle dose 5) and 2 participants will receive placebo.
  Participants in this Cohort will return for a second Treatment Period after a minimum washout period of 7 to 14 days. All 6 subjects will receive an inhaled dose of AZD8154 (large particle size).
  Interventions: Drug: AZD8154
- SAD Cohort 6 (Part 1) (Experimental): 6 Participants will receive AZD8154 (single inhaled small particle dose 6) and 2 participants will receive placebo.
  Interventions: Drug: AZD8154
- Cohort 1 (Part 2) (Experimental): All participants in this cohort will receive single IV dose of AZD8154 in Treatment Period 1 and then after washout period, will receive inhaled AZD8154 (small particle size) in Treatment Period 2.
  Interventions: Drug: AZD8154
- MAD Cohort 1 (Part 3) (Experimental): 6 Participants will receive AZD8154 (single inhaled dose 8) and 2 participants will receive placebo on Day 1. Participants will then receive multiple dosing of AZD8154 (inhaled dose 8) or placebo once daily from Day 4 to Day 12.
  Interventions: Drug: AZD8154
- MAD Cohort 2 (Part 3) (Experimental): 6 Participants will receive AZD8154 (single inhaled dose 9) and 2 participants will receive placebo on Day 1. Participants will then receive multiple dosing of AZD8154 (Inhaled dose 9) or placebo once daily from Day 4 to Day 12.
  Interventions: Drug: AZD8154
- MAD Cohort 3 (Part 3) (Experimental): 6 Participants will receive AZD8154 (single inhaled dose 10) and 2 participants will receive placebo on Day 1. Participants will then receive multiple dosing of AZD8154 (inhaled dose 10) or placebo once daily from Day 4 to Day 12.
  Interventions: Drug: AZD8154

INTERVENTIONS:
Drug: AZD8154 — SAD Part 1; 6 cohorts which receive single dosing. One cohort is invited back for large particle administration. Part 2; 1 cohort which receives IV dose and then inhaled administration of AZD8154. MAD Part 3; 3 cohorts will receive inhaled multiple dosing. Additional doses are provisional and could be adjusted based on the emerging data from the previous dose by the safety review committee (SRC).

SUMMARY:
This study is a Phase 1, first in human (FiH) study, consisting of 3 parts (Part 1, Part 2, and Part 3) in healthy male and female participants of non-childbearing potential, performed at a single study center. Part 1 of this study will be a randomized, single-blind, placebo-controlled, single ascending dose (SAD) in healthy male and female participants of non-childbearing potential. Six dose levels of AZD8154 are planned to be investigated. Depending on emerging data, 1 to 2 additional dose levels may be added at the discretion of the Sponsor. Furthermore, one dose level will be repeated using the same formulation of AZD8154 but with a larger particle size (Part 1 only). Part 2 of this study will be a single cohort, open-label, 2-period, study to compare a single inhaled dose of AZD8154 (small particle size) nebuliser suspension with a single IV dose of AZD8154. Part 3 will be a single blind placebo controlled, multiple ascending doses (MAD) sequential design study in healthy male and/or female subjects of non childbearing potential conducted at a single center. Part 3:Three (3) inhaled dose levels of AZD8154 are planned to be investigated. Depending on the emerging data, up to 2 additional inhaled dose levels may be added at the discretion of the Sponsor.

DETAILED DESCRIPTION:
This is a phase 1 study to assess the safety, tolerability and pharmacokinetics of AZD8154 following single and multiple ascending dose administration in healthy participants. This study will have 3 parts (Part 1, Part 2, and Part 3). Part 1 consists of six cohorts, each consisting of 8 participants. Depending on emerging PK and adverse event (AE) data, 1 to 2 additional inhaled dose levels, within the pre-specified dose range, may be added at the discretion of the Sponsor. One dose level cohort selected based on emerging data will be repeated using the same formulation of AZD8154 but with a larger particle size. The selected cohort (e.g., Cohort 5), referred to as the "Large Particle Size Cohort", will be dosed at the same dose level with a larger particle size after a minimum washout period of 7 to 14 days between each dose administration.

Small Particle Size Cohorts:

Within each cohort, 6 participants will be randomized to receive an inhaled dose of AZD8154 (small particle size) and 2 participants will be randomized to receive inhaled placebo. Dosing for each ascending dose cohort will proceed with 2 participants in a sentinel cohort, such that 1 participant will be randomized to receive placebo and 1 participant will be randomized to receive AZD8154 (small particle size).

Large Particle Size Cohort:

For the selected Large Particle Size Cohort, the 6 participants that received AZD8154 (small particle size) will return for a second Treatment Period after a minimum washout period of 7 to 14 days. All 6 participants will receive an inhaled dose of AZD8154 (large particle size), at the same dose level that they received AZD8154 (small particle size) in Treatment Period 1. The duration of the washout period is based on the predicted half-life of AZD8154 and was selected to diminish the impact of carry-over effects from the first Treatment Period.

Part 2: Part 2 of this study will be a single cohort. One cohort consisting of 6 participants will be enrolled into Part 2 of the study. All subjects will receive AZD8154 IV in Treatment Period 1 and then after washout, receive inhaled AZD8154 (small particle size) in Treatment Period 2. Intravenous dosing will proceed with 1 participant in a sentinel cohort, no sentinel dosing will be done in the inhaled dosing period.

Part 3: Three cohorts (MAD Cohort 1 to Cohort 3), each consisting of 8 participants, will participate in Part 3 of the study. Within each cohort, 6 participants will be randomized to receive an inhaled dose of AZD8154 and 2 participants will be randomized to receive inhaled placebo. Dosing for each ascending dose cohort will proceed with 2 participants in a sentinel cohort, such that 1 participant will be randomized to receive placebo and 1 participant will be randomized to receive AZD8154. In Part 3, participants will be randomized to receive an inhaled dose of AZD8154 nebuliser suspension or placebo. Three (3) inhaled dose levels of AZD8154 that are administered once daily are planned to be investigated. Based upon emerging PK and safety data in MAD Cohorts 1 to 3, up to 2 additional inhaled dose levels, within the pre-specified dose range, may also be added at the discretion of the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent before any study specific procedures.
2. Healthy male and/or female participants of non-childbearing potential aged 18 to 45 years (inclusive at the Screening Visit) with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit, must not be lactating and must be of non-child-bearing potential, confirmed at Screening by fulfilling one of the following criteria: 3.1. Postmenopausal defined as amenorrhea for at least 12 months or more following cessation of all exogenous hormonal treatments and Follicle-stimulating hormone (FSH) levels in the postmenopausal range. 3.2. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
4. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive, and weigh at least 60 kg and no more than 100 kg inclusive.
5. Subject has a FEV1 ≥ 80% of the predicted value regarding age, height, gender and ethnicity at the Screening Visit.

Exclusion Criteria:

1. History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. Subject is immuno-compromised.
3. History of diabetes, impaired fasting glucose, metabolic syndrome, hypertriglyceridemia or familial lipid disorders.
4. Current or previous history of malignancy of any kind except cutaneous basal or squamous cell carcinoma successful treated with therapy.
5. History of any respiratory disorders such as asthma, chronic obstructive pulmonary disease (COPD) or idiopathic pulmonary fibrosis (IPF).
6. Subject with latent or active tuberculosis (TB), as conformed by a positive QuantiFERON® - TB Gold test or as judged by the Investigator at the Screening Visit.
7. History or presence of GI, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs, or bowel disorders not otherwise specified.
8. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the (first) administration of the IMP.
9. Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results, defined as the following:

   9.1. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > the upper limit of the normal (ULN) laboratory range.

   9.2. Bilirubin > 1.5 times the ULN laboratory range. 9.3. Absolute neutrophil count < lower limit of normal (LLN). 9.4. Absolute lymphocyte count < LLN. 9.5. Fasting plasma glucose > ULN. 9.6. Triglycerides > ULN.
10. Any positive result at the Screening Visit for serum hepatitis B surface antigen (HBsAg) OR hepatitis B core antibodies (anti-HBc), hepatitis C antibody and human immunodeficiency virus (HIV).
11. Abnormal vital signs, after 5 minutes supine rest, defined as any of the following:

    11.1. Systolic BP < 90 mmHg or > 140 mmHg. 11.2. Diastolic BP < 50 mmHg or > 90 mmHg. 11.3. Heart rate < 50 or > 90 beats per minute (bpm).
12. Any clinically important abnormalities in rhythm, conduction or morphology of the 12-lead safety and any clinically important abnormalities in the 12-Lead dECG as considered by the Investigator that may interfere with the interpretation of QT interval corrected for heart rate using Fridericia's formula (QTcF) interval changes, including abnormal ST-T-wave morphology, particularly in the CSP defined primary lead for dECG analysis or left ventricular hypertrophy.

    12.1. Prolonged QTcF > 450 ms or shortened QTcF < 340 ms or family history of long QT syndrome.

    12.2. PR (PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation).

    12.3. PR (PQ) interval prolongation (> 220 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree atrioventricular (AV) block, or AV dissociation.

    12.4. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. participants with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of e.g., ventricular hypertrophy or pre-excitation.
13. Previous use of a mechanistic target of rapamycin (mTOR) antagonist (e.g., rapamycin, everolimus) or PI3K inhibitor (selective or non-selective PI3K inhibitors).
14. Known or suspected history of drug abuse as judged by the Investigator.
15. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the previous 3 months.
16. History of alcohol abuse or excessive intake of alcohol as judged by the Investigator.
17. Positive screen for drugs of abuse or cotinine (nicotine) at the Screening Visit or admission to the Clinical Unit or positive screen for alcohol on admission to the Clinical Unit before the (first) administration of the IMP.
18. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD8154.
19. Receipt of live attenuated vaccines 2 months before (first) administration of the IMP and 3 months after the last IMP administration.
20. Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate) as judged by the Investigator.
21. Use of drugs with CYP3A enzyme inducing or inhibition properties such as St John's Wort within 3 weeks before (first) administration of IMP.
22. Use of any prescribed or nonprescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks before the (first) administration of the IMP or longer if the medication has a long half-life.
23. Plasma donation within 1 month of the Screening Visit or any blood donation/blood loss > 500 mL during the 2 months before the Screening Visit.
24. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the (first) administration the IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest. Note: participants consented and screened, but not randomized in this study or a previous Phase 1 study, are not excluded.
25. Involvement of any Astra Zeneca or study site employee or their close relatives.
26. Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the Screening Period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
27. Participants who cannot communicate reliably with the Investigator and/or is not able to read speak and understand German language.
28. Vulnerable participants, e.g., kept in detention, protected adults under guardianship, trusteeship or committed to an institution by governmental or juridical order.

    In addition, any of the following is regarded as a criterion for exclusion from the genetic research:
29. Previous bone marrow transplant.
30. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (Part 1 & 2) | From Day-1 up to follow-up visit (6 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses; inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with adverse events (Part 3) | From Day-1 up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal findings in 12-lead digital electrocardiography (ECG) (Part 1) | At Treatment period (Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
Number of participants with abnormal findings in 12-lead digital ECG (Part 2) | At Treatment Periods 1 and 2 (Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal findings in 12-lead digital ECG (Part 3) | At Treatment period (Days 1 to 15).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal pulse rate (Part 1) | From screening up to the treatment period (Day -1, Days 1 to 3)
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
Number of participants with abnormal pulse rate (Part 2) | From screening (Days -28 to -2) up to follow-up visit (6 ± 1 days post-dose)
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal pulse rate (Part 3) | From screening (Days-28 to -2) up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal findings in telemetry (Part 1) | At Treatment Period (Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
Number of participants with abnormal findings in telemetry (Part 2) | At Treatment Periods 1 (Days 1 to 3) and 2 (Days 1 to 3 and Day 4).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal findings in telemetry (Part 3) | At Treatment Period (Days 1 to 15)
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal hematology (Part 1 & Part 2) | From screening up to Treatment Period (Day-1, Days 1 to 3).
  To assess white blood cell count (WBC), red blood cell count (RBC), neutrophils absolute count, lymphocytes absolute count, monocytes absolute count, eosinophils absolute count, basophils absolute count as a variable of safety and tolerability of AZD8154 following inhaled administration of single ascending doses and inhaled and intravenous (IV) administration of single doses to healthy participants to healthy participants.
Number of participants with abnormal hematology (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess white blood cell count (WBC), red blood cell count (RBC), neutrophils absolute count, lymphocytes absolute count, monocytes absolute count, eosinophils absolute count, basophils absolute count the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal blood pressure (systolic and diastolic) (Part 1 & Part 2) | From screening up to the treatment period (Day -1, Days 1 to 3)
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses and inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal blood pressure (systolic and diastolic) (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal findings in respiratory rate (Part 1) | From screening up to the treatment period (Day -1, Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
Number of participants with abnormal findings in respiratory rate (Part 2) | From screening up to follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal findings in respiratory rate (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal physical examination (Part 1) | From screening up to follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants. The brief physical examinations will include an assessment of the general appearance, skin, cardiovascular system, respiratory and abdomen.
Number of participants with abnormal physical examination (Part 2) | From screening up to follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants. The brief physical examinations will include an assessment of the general appearance, skin, cardiovascular system, respiratory and abdomen.
Number of participants with abnormal physical examination (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy subjects. The brief physical examinations will include an assessment of the general appearance, skin, cardiovascular system, respiratory and abdomen.
Number of participants with abnormal findings in oral body temperature (Part 1) | From screening up to Treatment period (Day -1, Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
Number of participants with abnormal findings in oral body temperature (Part 2) | From screening up to Treatment Periods 1 and 2.
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal findings in oral body temperature (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Forced expiratory volume in 1 second (FEV1) (Part 1) | At Days-28 to -2, Day -1, Days 1 to 3.
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
FEV1 (Part 2) | At Days-28 to -2, Day -1, Days 1 to 3, and follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
FEV1 (Part 3) | At Days-28 to -2, Day -1, Days 1 to 12, and follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Forced vital capacity (FVC) (Part 1) | At Days-28 to -2, Day -1, Days 1 to 3.
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
FVC (Part 2) | At Days-28 to -2, Day -1, Days 1 to 3, and follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
FVC (Part 3) | At Days-28 to -2, Day -1, Days 1 to 12, and follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal electrolytes (Part 1) | From screening up to Treatment Period (Day-1, Days 1 to 3).
  To assess serum level of sodium, potassium, calcium, and phosphate as a variable of safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
Number of participants with abnormal electrolytes (Part 2) | From screening up to follow-up visit (6 ± 1 days post-dose).
  To assess serum level of sodium, potassium, calcium, and phosphate as a variable of safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal electrolytes (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess serum level of sodium, potassium, calcium, and phosphate as a variable of safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal hemoglobin (Hb) (Part 1) | From screening up to Treatment Period (Day-1, Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
Number of participants with abnormal hemoglobin (Hb) (Part 2) | From screening up to follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal hemoglobin (Hb) (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal hematocrit (Part 1) | From screening up to Treatment Period (Day-1, Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
Number of participants with abnormal hematocrit (Part 2) | From screening up to follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal hematocrit (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal mean corpuscular volume (MCV) (Part 1) | From screening up to Treatment Period (Day-1, Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
Number of participants with abnormal mean corpuscular volume (MCV) (Part 2) | From screening up to follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal mean corpuscular volume (MCV) (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal mean corpuscular hemoglobin (MCH) (Part 1) | From screening up to Treatment Period (Day-1, Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
Number of participants with abnormal mean corpuscular hemoglobin (MCH) (Part 2) | From screening up to follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal mean corpuscular hemoglobin (MCH) (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal mean corpuscular hemoglobin concentration (MCHC) (Part 1) | From screening up to Treatment Period (Day-1, Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
Number of participants with abnormal mean corpuscular hemoglobin concentration (MCHC) (Part 2) | From screening up to follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal mean corpuscular hemoglobin concentration (MCHC) (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal platelet count (Part 1) | From screening up to Treatment Period (Day-1, Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
Number of participants with abnormal platelet count (Part 2) | From screening up to follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal platelet count (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Number of participants with abnormal reticulocytes absolute count (Part 1) | From screening up to Treatment Period (Day-1, Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants.
Number of participants with abnormal reticulocytes absolute count (Part 2) | From screening up to follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants.
Number of participants with abnormal reticulocytes absolute count (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy participants.
Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) (Part 1 & Part 2) | At Day -1, Days1 to 3 and follow-up visit (6 ± 1 days post-dose).
  The DLCO assessment will be performed in Part 1 of the study. The DLCO assessments will be performed in Part 2, only if emerging data in Part 1 indicates that it is needed. The DLCO should be performed according to the American thoracic society (ATS)/ European respiratory society (ERS) guidelines. Post dose DLCO will only be performed if a reduction is observed in FEV1 or FVC (≥ 12%) starting 6 hours after IMP administration.
Diffusing Capacity of the Lungs for Carbon Monoxide (DLCO) (Part 3) | At Day -1, Days 1 to 12, and follow-up visit (7-10 days post final dose).
  The DLCO assessments will be performed in Part 2 and Part 3, only if emerging data in Part 1 indicates that it is needed. The DLCO should be performed according to the ATS/ERS guidelines. Post dose DLCO will only be performed if a reduction is observed in FEV1 or FVC (≥ 12%) starting 6 hours after IMP administration.
Number of participants with abnormal clinical chemistry (Part 1) | From screening up to Treatment Period (Day-1, Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants. The laboratory variables to be measured are: total bilirubin, unconjugated bilirubin, thyroxine (T4), thyroid stimulating hormone (TSH), triglycerides, follicle stimulating hormone (FSH), creatinine, albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), cystatin C, gamma glutamyl transpeptidase, and urea.
Number of participants with abnormal clinical chemistry (Part 2) | From screening up to follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants. The laboratory variables to be measured are: total bilirubin, unconjugated bilirubin, thyroxine (T4), thyroid stimulating hormone (TSH), triglycerides, follicle stimulating hormone (FSH), creatinine, albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), cystatin C, gamma glutamyl transpeptidase, and urea.
Number of participants with abnormal clinical chemistry (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy subjects. The laboratory variables to be measured are: total bilirubin, unconjugated bilirubin, thyroxine (T4), thyroid stimulating hormone (TSH), triglycerides, follicle stimulating hormone (FSH), creatinine, albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), cystatin C, gamma glutamyl transpeptidase, and urea.
Number of participants with abnormal urinalysis (Part 1) | From screening up to Treatment Period (Day-1, Days 1 to 3).
  To assess the safety and tolerability of AZD8154 following inhaled administration of single ascending doses to healthy participants. The laboratory variables to be measured are: protein, glucose, and blood.
Number of participants with abnormal urinalysis (Part 2) | From screening up to follow-up visit (6 ± 1 days post-dose).
  To assess the safety and tolerability of AZD8154 following inhaled and intravenous (IV) administration of single doses to healthy participants. The laboratory variables to be measured are: protein, glucose, and blood.
Number of participants with abnormal urinalysis (Part 3) | From screening up to follow-up visit (7-10 days post final dose).
  To assess the safety and tolerability of AZD8154 following inhaled administration of multiple ascending doses to steady state to healthy subjects. The laboratory variables to be measured are: protein, glucose, and blood.

SECONDARY OUTCOMES:
Observed maximum plasma concentration (Cmax) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the Cmax of AZD8154 following inhaled administration of single ascending doses and intravenous (IV) doses of AZD8154 in healthy participants and to study the influence of particle size on AZD8154 PK parameters, to assess the time required to reach steady state, the degree of accumulation and the time dependency of the pharmacokinetics.
Time to reach peak or maximum observed concentration or response following drug administration (tmax) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the tmax of AZD8154 following inhaled administration of single ascending doses, IV doses of AZD8154, inhaled administration of single doses in healthy participants, and to study the influence of particle size on AZD8154 PK parameters.
Terminal elimination rate constant (λz) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the λz of AZD8154 following inhaled and IV doses of AZD8154, inhaled administration of single doses in healthy participants, and to study the influence of particle size on AZD8154 PK parameters.
Half life associated with terminal slope (λz) of a semi logarithmic concentration time curve (t½λz) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the t½λz of AZD8154 following inhaled administration of single ascending doses, IV doses of AZD8154, inhaled administration of single doses in healthy participants, and to study the influence of particle size on AZD8154 PK parameters.
Area under the plasma concentration time curve from time zero to 24 hours after dosing (AUC(0 24)) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the AUC(0 24) of AZD8154 following inhaled administration of single ascending doses, inhaled administration of single doses in healthy participants, and to study the influence of particle size on AZD8154 PK parameters.
Area under the plasma concentration curve from time zero to the time of last quantifiable analyte concentration (AUClast) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the AUClast of AZD8154 following inhaled administration of single ascending doses and IV doses of AZD8154, inhaled administration of single doses in healthy participants, and to study the influence of particle size on AZD8154 PK parameters.
Area under plasma concentration time curve from time zero extrapolated to infinity (AUC) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the AUC of AZD8154 following inhaled administration of single ascending doses and IV doses of AZD8154, inhaled administration of single doses in healthy participants, and to study the influence of particle size on AZD8154 PK parameters.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the CL/F of AZD8154 following inhaled administration of single ascending doses, inhaled administration of single doses in healthy participants, and to study the influence of particle size on AZD8154 PK parameters.
Mean residence time of the unchanged drug in the systemic circulation (MRT) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the MRT of AZD8154 following inhaled administration of single ascending doses and IV doses of AZD8154, inhaled administration of single doses in healthy participants, and to study the influence of particle size on AZD8154 PK parameters.
Volume of distribution at terminal phase (intravenous dosing) (Vz) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the Vz of AZD8154 following IV administration.
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the Vz/F of AZD8154 following inhaled administration of single ascending doses, inhaled administration of single doses in healthy participants, and to study the influence of particle size on AZD8154 PK parameters.
Area under the plasma concentration time curve from time zero to time of last quantifiable analyte concentration divided by the dose administered (AUClast/D) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the AUClast/D of AZD8154 following inhaled administration of single ascending doses, inhaled administration of single doses in healthy participants, and to study the influence of particle size on AZD8154 PK parameters.
Area under the plasma concentration time curve from time zero extrapolated to infinity divided by the dose administered (AUC/D) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the AUC/D of AZD8154 following inhaled administration of single ascending doses, inhaled administration of single doses in healthy participants, and to study the influence of particle size on AZD8154 PK parameters.
Observed maximum plasma concentration divided by the dose administered (Cmax/D) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the Cmax/D of AZD8154 following inhaled administration of single ascending doses, inhaled administration of single doses in healthy participants, and to study the influence of particle size on AZD8154 PK parameters.
Time of last quantifiable plasma concentration (tlast) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the tlast of AZD8154 following inhaled administration of single ascending doses, inhaled administration of single doses in healthy participants, and to study the influence of particle size on AZD8154 PK parameters.
Total body clearance of drug from plasma after intravascular administration (CL) | At treatment period [Days 1 to 3]
  To assess the CL of AZD8154 following IV doses of AZD8154.
Volume of distribution at steady state from a systemic dose (Vss) | At treatment period [Days 1 to 3]
  To assess the Vss of AZD8154 following IV doses of AZD8154.
Terminal half-life (t½) | At treatment period [Days 1 to 3]
  To assess the t½ of AZD8154 following IV doses of AZD8154.
Area under the plasma concentration time curve from time zero to 24 hours after dosing divided by the dose administered (AUC(0 24)/D) | At treatment period [Days 1 to 3 (Part 1 & 2)], Day 4 (Part 2) and [Days 1 to 12 (Part 3)]
  To assess the AUC (0-24)/D of AZD8154 following inhaled administration of single ascending doses of AZD8154, inhaled doses of AZD8154, to study the influence of particle size on AZD8154 PK parameters, and to assess the time required to reach steady state, the degree of accumulation and the time dependency of the pharmacokinetics.
Area under the concentration time curve in the dose interval (AUCτ) | At treatment period Days 1 to 12
  To assess the AUCτ of AZD8154 following multiple dose pharmacokinetics of AZD8154 and to assess the time required to reach steady state, the degree of accumulation and the time dependency of the pharmacokinetics.
Area under the concentration time curve in the dose interval divided by the dose administered (AUCτ/D) | At treatment period Days 1 to 12
  To assess the AUCτ/D of AZD8154 following multiple dose pharmacokinetics of AZD8154 and to assess the time required to reach steady state, the degree of accumulation and the time dependency of the pharmacokinetics.
Accumulation ratio based on AUCτ (Rac (AUC)) | At treatment period Days 1 to 12
  To assess the Rac (AUC) of AZD8154 following multiple dose pharmacokinetics of AZD8154 and to assess the time required to reach steady state, the degree of accumulation and the time dependency of the pharmacokinetics.
Accumulation ratio based on Cmax (Rac (Cmax)) | At treatment period Days 1 to 12
  To assess the Rac (Cmax) of AZD8154 following multiple dose pharmacokinetics of AZD8154 and to assess the time required to reach steady state, the degree of accumulation and the time dependency of the pharmacokinetics.
Temporal change parameter in systemic exposure [TCP (AUC)] | At treatment period Days 1 to 12
  To assess the TCP (AUC) of AZD8154 following multiple dose pharmacokinetics of AZD8154 and to assess the time required to reach steady state, the degree of accumulation and the time dependency of the pharmacokinetics.
Change from baseline concentration of 4 β hydroxy cholesterol | Change from baseline
  To assess the induction potential of AZD8154 on cytochrome P450 (CYP)3A by measuring 4 β hydroxy cholesterol at baseline and at steady state.
Mean absorption time (MAT) | At treatment period [Days 1 to 3 & Day 4]
  To assess MAT of AZD8154 following inhaled doses of AZD8154.
Fraction of administered dose systemically available (F) | At treatment period [Days 1 to 3 & Day 4]
  To assess F of AZD8154 following inhaled doses of AZD8154.

CONTACTS AND LOCATIONS:
Overall Officials: med. Rainard Fuhr, Dr, Principal Investigator — PAREXEL Early Phase Clinical Unit Berlin
Locations (1):
- Research Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No